CLINICAL TRIAL: NCT03333733
Title: Cluster Randomised Controlled Feasibility Study of HENRY; a Community Based Intervention Aimed at Reducing School Entry Obesity Rates
Brief Title: Protocol Feasibility Study of HENRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: NatCen Social Research (Unknown)
Responsible Party: Principal Investigator, Maria Bryant, Portfolio lead for Diet, Obesity and Lifestyle, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDF-2014-07-052
Record Dates: First submitted 2017-09-28; First posted 2017-11-07 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Childhood Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Health; Exercise; Nutritional Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Treatment allocation will be withheld from research staff collecting the data. Screening forms will not indicate whether they have been recruited from active or control Centres The chief investigator, trial coordinator and statistician will not be provided details of treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HENRY (Experimental): Children's Centres within local authorities that have been randomised to the experimental arm, HENRY, will receive staff training to deliver the training and be asked to implement at least two programmes per year. Parents enrolled to attend HENRY programmes will then be invited to take part in the research.
  Interventions: Behavioral: HENRY
- Waiting list control (No Intervention): Children's Centres within local authorities that have been randomised to the control arm will continue with usual practice. Parents attending another programme (Stay and Play) will be invited to take part in the research. At the end of the follow-up period, they will be offered training to deliver HENRY programmes although this will not be compulsory.

INTERVENTIONS:
Behavioral: HENRY — HENRY is an 8-week programme delivered in Children's Centres, aiming to provide parents with skills and knowledge to support healthy lifestyles in preschool children and their families. It is currently delivered in ~ 35 local areas across England and Wales by trained health and community practitioners. Training includes:
  Centre Level Training: to equip staff with knowledge and skills to promote and provide healthy nutrition within early years settings and support parents to provide healthy family lifestyles and nutrition for their families. The theoretical underpinning combines proven models of behaviour change including the Family Partnership Model, motivational interviewing and solution-focused support.
  Practitioner Level Training: to deliver the 8-week HENRY programme, which aims to build parents' skills, knowledge and confidence to change old habits and provide healthier nutrition for their young children.
  Other Names: Health, Exercise, Nutrition for the Really Young
  Arms: HENRY

SUMMARY:
Tackling obesity is a public health priority. Childhood obesity is of particular concern due to its impact on physiological and psychological health and likelihood of tracking into adulthood, with associated diseases and disorders and financial burden to the NHS. Once established, obesity is hard to treat. Therefore, prevention strategies aimed at children are essential.

This study aims to determine the feasibility of undertaking a full trial to evaluate the clinical effectiveness of the HENRY (Health, Exercise, Nutrition for the Really Young) programme in preventing childhood obesity. It is a multi-centre, open labelled, two group, prospective, cluster randomised, controlled, feasibility study aiming to recruit 120 parents from 12 Children's Centres.

HENRY (Health, Exercise, Nutrition for the Really Young) is an 8 week community based intervention delivered in settings such as Children's Centres, aimed at preventing childhood obesity by supporting families to make positive lifestyle changes. It is currently widely delivered across the UK. Preliminary data indicates that HENRY may be effective at reducing childhood obesity and improving family health, although a robust evaluation has not yet been conducted. A good deal of public money has already been used to develop and commission HENRY and it is essential to demonstrate clear benefits of the programme before further funding. This study will determine whether a definitive randomised controlled trial (RCT) of HENRY is feasible. 12 Children's Centres will be recruited from two local authorities. From these, half will be randomised to deliver HENRY programmes.

From the participating Children's Centres, 120 parents will be recruited. All participants will be asked to meet with a researcher twice in their home, 12 months apart. During the visit, parents will complete 4 questionnaires around diet and lifestyle. Height and weight measurements will also be taken from the parent (optional) and child (compulsory). The decision of whether a RCT is feasible will be based on whether it is possible to recruit local authorities, children's centres and parents to take part; ensure staff can be adequately trained to deliver programmes within specified timeframes; and whether proposed data can be adequately gathered.

DETAILED DESCRIPTION:
Background:

Childhood obesity impacts physiological and psychological health that tracks into adulthood; increasing risk of morbidity and mortality [1, 2]. It incurs significant costs on the UK economy, with an expected 7-fold increase in related NHS costs by 2020, and forecasted £2 billion annual spend by 2030[3]. Tackling obesity is a key NHS public health priority, with government strategies aimed at reversing the trend of rising childhood obesity levels to return to those of 2000. Whilst treating obesity remains a priority, there are compelling arguments to prevent its onset. Establishing healthy behaviours in early childhood is critical for optimum growth and development [4]. Further, poor eating patterns developed early can persist and are associated with chronic diseases in adulthood (e.g. cardiovascular disease, type-2-diabetes [5]). Once established, obesity is difficult to reverse[6]; strengthening the case for primary prevention[7]. Early preventive interventions are therefore essential to impact the health of our children now and in the future [8].

Interventions aimed at treating obesity report inconsistent results [9-11, 6, 12, 13], though there is agreement that multi-component interventions, especially those engaging parents have a greater impact [14, 6]. Proposed research involves an independent evaluation of an existing preschool obesity prevention intervention. The HENRY programme was developed in 2007 with Department of Health and Department for Education support and is currently delivered across the UK by approximately 35 Local Authorities providing ~190 courses/year. Over 10,000 families have already participated. It is delivered in the community, predominantly by Children's Centre staff [15]. HENRY uses a responsive approach to provide practical guidance and improve parenting skills, aimed at enhancing family homes and Children's Centre environments. These are intervention targets that are consistent with recent literature in childhood obesity. Preliminary data indicates that HENRY may be effective at reducing childhood obesity and improving family health [15] although evidence to date has not compared findings with parents who have not attended HENRY; thus, further robust evaluation using a RCT design is needed to confirm its effectiveness. A good deal of public money has already been used to develop and commission HENRY and it is essential to demonstrate clear benefits of the programme before further funding. Given the uncertainties associated with recruiting local authorities, service providers and Children's Centres, it is necessary to conduct research in advance of a definitive multi-site trial. The models of commissioning and delivering HENRY are complex and vary by location. In some instance, HENRY is commissioned by local authorities and delivered by existing Centre staff. In others, Children's Centres are tendered to external service providers (e.g. Barnardo's) who are responsible for commissioning programmes such as HENRY. This study will assess feasibility of the planned recruitment rate at the authority, Centre and parent level and ensure competence of programme delivery; in addition to providing vital information for calculation of the sample size for the future trial. A future trial will be used to offer commissioners an evidence based intervention, tested in Children's Centres in the UK and to provide much needed evidence on the effectiveness of early obesity prevention in primary care settings.

Aim:

The feasibility study aims to determine the feasibility of undertaking a full trial to evaluate the clinical effectiveness of the HENRY programme in preventing childhood obesity.

Primary Objectives:

1. To determine whether it is feasible to recruit local authorities/service providers that are willing to nominate Children's Centres to be involved in the research (allowing randomisation where they would usually select Centres most in need).
2. To assess the time required to train and certify staff to delivery HENRY programmes in order to propose a clear process and timeline for the definitive trial
3. To determine whether it is possible to recruit parents to the study, who are enrolled to attend a HENRY programme; and the practicality of recruiting parents to the study from control Centres, where the pathway to recruitment is less defined compared to the HENRY Centres.
4. To explore the current landscape of HENRY commissioning, provision and delivery via postal screening questionnaire and qualitative data collection in areas currently delivering HENRY
5. To explore the level of contamination, including the degree to which parents use multiple Centres, the amount of contamination through social networks (control and HENRY parents sharing knowledge) and the possibility of HENRY trained facilitators sharing knowledge within control Centres.

Secondary Objectives:

1. To examine the acceptability and completeness of the proposed methods of data collection to ensure they are feasible for the definitive trial.
2. To gather data to allow estimation of the sample size requirements for the definitive trial.
3. To assess the acceptability of the design for parents, commissioners and Centre staff; particularly related to withholding HENRY training in control Centres until the end of the study.
4. To provide evidence that participants fully understand and accept their involvement in the study via feedback questionnaire and qualitative assessment.

4. To determine the practicalities of delivering the required number of HENRY programmes within the trial period in regards to programme implementation.

Progression rules:

1. Recruitment of local authorities (and their service providers (if applicable)): Green = two local authorities within 12 months; Red = Less than two local authorities within 12 months
2. Randomisation of Children's Centres: Green = at least 12 Centres randomised within 12 months; Amber = 9-12 Centres randomised within 12 months; Red = less than 9 randomised within 12 months.
3. Recruitment of parents: Green = an average of at least 4 parents registered per programme (or control group equivalent); Amber = 3 parents registered per programme; Red = less than 3 parents registered per programme.

Objectives related to staff training, collection of data and estimating sample size are included to support the design of the definitive trial, rather than acting as progression criteria.

Design:

This is a multi-centre, open labelled, two group, prospective, cluster randomised, controlled, feasibility study aiming to recruit 120 parents from 12 Children's Centres. Cluster randomisation has been chosen to reduce between-group contamination as HENRY is a group-based intervention which aims to provide practical guidance and improve parenting skills, intended at enhancing family homes and Children's Centre environments. All parents registered from HENRY Centres will receive the intervention and therefore it is not possible to use parents as the unit of randomisation. Centres and participants will, of necessity, be aware of treatment allocation but collection of outcomes will be performed by researchers blind to treatment allocation. Randomisation of Children's Centres will be performed by the statistician at the Clinical Trials Research Unit (CTRU).

Within each of the two local authorities, three Centres will be randomised to HENRY and three will be randomised to the control arm (training to deliver the HENRY programme in these Centres will not occur until the end of the study). Historically, when HENRY is commissioned by an area, it is the local authority which determines which Centre's will receive the intervention. In areas where HENRY is provided by external partners (e.g. Banardos), this is determined by the service provider. To maintain some autonomy by the commissioners, local authorities/service providers will be asked to allow randomisation of half of the Centres they propose to the intervention and half to the control arm. Additional training will be offered to those in the wait list control group after follow-up data have been collected (although attendance will not be compulsory).

Screening of parents will take place at Children's Centres by Centre staff and during telephone calls from NatCen (an independent social research agency (http://natcen.ac.uk) that have no role in delivery of the intervention). Consent and recruitment will occur in parent's homes and will be undertaken by staff from NatCen. Self-report questionnaires at 12 months will be collected by NatCen researchers within family homes, or at the Children's Centre if preferred by the parent. Engagement with the intervention will be assessed by an independent member of the trial team at approximately three and six months. Contamination will be assessed using a combination of quantitative (e.g. data on facilitators working in multiple Centres) and qualitative (e.g. parent focus groups) measures by mapping intervention components against their potential to impact on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* SITE level Local authorities (or other associations that commission HENRY in Children's Centres), Children's Centres and parents meeting all of the relevant inclusion criteria, and none of the relevant exclusion criteria, will be considered for participation in the study.

Local authorities (and service providers if applicable):

* Local Authorities must nominate a minimum of 6 Children's Centres and formally agree to allow randomisation of the Centres. Where possible, Centres should be in geographically separate areas to protect against contamination (judged on a case by case basis). Local authorities using external teams outside of the Centre to deliver HENRY programmes (e.g. health visitors) will be eligible, in addition to those wishing to train internal Centre staff to deliver programmes (the most common model currently used).
* Included local authorities may be completely new to HENRY (having never trained or delivered HENRY) or contain at least 6 Centres that are within HENRY 'naïve' clusters. Clusters are defined as a number of Children's Centres that are close to each other or grouped for management purposes. HENRY naive clusters are:
* A group of Centres within a cluster that do not include any Centres that are (a) currently delivering HENRY or (b) have been trained to, or delivered HENRY within the past 2 years.

PARENT level The target population for the intervention are parents of preschool children; mothers, fathers and carers (e.g. with children living in stable /long-term foster care).

* Parents must have at least 1 child aged 6 months - 5 years (18 months-6 years at follow-up). If more than one child in the family fulfils eligibility criteria, the youngest child (by birth timing if twins) will be considered as the reference child (from which data will be collected).
* Parents must be willing to attend the programme sessions (intervention Centres) and willing to provide data in accordance with the data collection protocol. Parents will be provided with full details of the data collection requirements in advance so that they can make informed decisions as to whether to participate.
* Parents must speak English, unless they wish to bring their own interpreter with them (e.g. family member) (the intervention and data collection forms are currently only available in English).

Exclusion Criteria:

* - SITE level

  * Children's Centres that have delivered HENRY programmes within the last 2 years or where staff have received HENRY training within the last 2 years.

PARENT level

* Parents with severe learning difficulties that preclude them taking part in group sessions in which they need to be able to read and write, judged on a case by case basis with consultation with the HENRY team where appropriate.
* Parents whose reference child is tube fed (PEG or nasogastric) or with other known clinical conditions likely to affect growth over the period of the trial (e.g. cancer, coeliac disease, or renal or cardiac problems). A detailed list of excluded conditions will be provided at screening, with any uncertainties resolved via clinical input from the HENRY team.
* Parents who have attended a HENRY group for a previous child.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-07-30 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Number of centres recruited | 12 months from ethical approval
Quality assurance in training achieved | 12 months from ethical approval
  Pass/fail of training completion recorded by central HENRY team
Number of parents recruited per centre | 12 months from completion of training
Intervention fidelity | 24 months from completion of training
  Adherence to manual identified through observations of intervention sessions
Contamination risk score | 24 months from completion of training
  Qualitatively assessed and assigned score. Combined risk probability and risk severity scores. Risk probability assessed with a 5-point ordinal scale, ranging from 1 (improbable frequency of risk) to 5 (frequent). Risk severity assessed with a 5-point ordinal scale ranging from A (severe likelihood that contamination will impact on the trial) to E (negligible impact). Combined responses mean that there are 25 possible responses with 5A representing greatest impact of contamination (Frequent and severe) to 1E (improbable contamination with negligible impact).

SECONDARY OUTCOMES:
Trial acceptability qualitatively assessed through interviews with participants | 24 months from centre recruitment
Reference child BMI z-score data | Measured at follow-up (12 months from parent recruitment)
  Effect size, variance and ICCs to determine sample size

OTHER OUTCOMES:
Reference child BMI z-score | Measured at baseline and follow-up (12 months from parent recruitment)
  Proposed definitive trial outcome - measured height/length and weight
Primary care giver BMI | Measured at baseline and follow-up (12 months from parent recruitment)
  Proposed definitive trial outcome - measured height and weight
Family eating activities | Measured at baseline and follow-up (12 months from parent recruitment)
  Proposed definitive trial outcome - 21-item Golan questionnaire
Parenting self-agency | Measured at baseline and follow-up (12 months from parent recruitment)
  Proposed definitive trial outcome - 5-item Dumka Parenting Self Agency Measure
Child feeding practices | Measured at baseline and follow-up (12 months from parent recruitment)
  Proposed definitive trial outcome -37-item Baughcum pre-schooler feeding questionnaire
Dental health | Measured at baseline and follow-up (12 months from parent recruitment)
  Proposed definitive trial outcome -6items related to tooth brushing, dental attendance and whether the child has received general anaesthetic treatment
Child activity/movement | Measured at baseline and follow-up (12 months from parent recruitment)
  Pedometer worn over 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine and Health, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh GK, Kogan MD, van Dyck PC. A multilevel analysis of state and regional disparities in childhood and adolescent obesity in the United States. J Community Health. 2008 Apr;33(2):90-102. doi: 10.1007/s10900-007-9071-7. PMID 18049885
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Wang YC, McPherson K, Marsh T, Gortmaker SL, Brown M. Health and economic burden of the projected obesity trends in the USA and the UK. Lancet. 2011 Aug 27;378(9793):815-25. doi: 10.1016/S0140-6736(11)60814-3. PMID 21872750
- [Background] Freedman DS, Dietz WH, Srinivasan SR, Berenson GS. The relation of overweight to cardiovascular risk factors among children and adolescents: the Bogalusa Heart Study. Pediatrics. 1999 Jun;103(6 Pt 1):1175-82. doi: 10.1542/peds.103.6.1175. PMID 10353925
- [Background] Oude Luttikhuis H, Baur L, Jansen H, Shrewsbury VA, O'Malley C, Stolk RP, Summerbell CD. Interventions for treating obesity in children. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD001872. doi: 10.1002/14651858.CD001872.pub2. PMID 19160202
- [Background] Waters E, de Silva-Sanigorski A, Hall BJ, Brown T, Campbell KJ, Gao Y, Armstrong R, Prosser L, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD001871. doi: 10.1002/14651858.CD001871.pub3. PMID 22161367
- [Background] Morandi A, Meyre D, Lobbens S, Kleinman K, Kaakinen M, Rifas-Shiman SL, Vatin V, Gaget S, Pouta A, Hartikainen AL, Laitinen J, Ruokonen A, Das S, Khan AA, Elliott P, Maffeis C, Gillman MW, Jarvelin MR, Froguel P. Estimation of newborn risk for child or adolescent obesity: lessons from longitudinal birth cohorts. PLoS One. 2012;7(11):e49919. doi: 10.1371/journal.pone.0049919. Epub 2012 Nov 28. PMID 23209618
- [Background] Leblanc ES, O'Connor E, Whitlock EP, Patnode CD, Kapka T. Effectiveness of primary care-relevant treatments for obesity in adults: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2011 Oct 4;155(7):434-47. doi: 10.7326/0003-4819-155-7-201110040-00006. PMID 21969342
- [Background] Loveman E, Frampton GK, Shepherd J, Picot J, Cooper K, Bryant J, Welch K, Clegg A. The clinical effectiveness and cost-effectiveness of long-term weight management schemes for adults: a systematic review. Health Technol Assess. 2011 Jan;15(2):1-182. doi: 10.3310/hta15020. PMID 21247515
- [Background] Summerbell CD, Ashton V, Campbell KJ, Edmunds L, Kelly S, Waters E. Interventions for treating obesity in children. Cochrane Database Syst Rev. 2003;(3):CD001872. doi: 10.1002/14651858.CD001872. PMID 12917914
- [Background] Blake-Lamb TL, Locks LM, Perkins ME, Woo Baidal JA, Cheng ER, Taveras EM. Interventions for Childhood Obesity in the First 1,000 Days A Systematic Review. Am J Prev Med. 2016 Jun;50(6):780-789. doi: 10.1016/j.amepre.2015.11.010. Epub 2016 Feb 22. PMID 26916260
- [Background] Redsell SA, Edmonds B, Swift JA, Siriwardena AN, Weng S, Nathan D, Glazebrook C. Systematic review of randomised controlled trials of interventions that aim to reduce the risk, either directly or indirectly, of overweight and obesity in infancy and early childhood. Matern Child Nutr. 2016 Jan;12(1):24-38. doi: 10.1111/mcn.12184. Epub 2015 Apr 20. PMID 25894857
- [Background] Hillier F, Pedley C, Summerbell C. Evidence base for primary prevention of obesity in children and adolescents. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2011 Mar;54(3):259-64. doi: 10.1007/s00103-010-1227-4. PMID 21347757
- [Background] Willis TA, George J, Hunt C, Roberts KP, Evans CE, Brown RE, Rudolf MC. Combating child obesity: impact of HENRY on parenting and family lifestyle. Pediatr Obes. 2014 Oct;9(5):339-50. doi: 10.1111/j.2047-6310.2013.00183.x. Epub 2013 Jul 2. PMID 23818487
- [Derived] Stamp E, Schofield H, Roberts VL, Burton W, Collinson M, Stevens J, Farrin A, Rutter H, Bryant M. Contamination within trials of community-based public health interventions: lessons from the HENRY feasibility study. Pilot Feasibility Stud. 2021 Mar 26;7(1):88. doi: 10.1186/s40814-021-00805-3. PMID 33771233
- [Derived] Bryant M, Collinson M, Burton W, Stamp E, Schofield H, Copsey B, Hartley S, Webb E, Farrin AJ. Cluster randomised controlled feasibility study of HENRY: a community-based intervention aimed at reducing obesity rates in preschool children. Pilot Feasibility Stud. 2021 Feb 26;7(1):59. doi: 10.1186/s40814-021-00798-z. PMID 33632330
- [Derived] Bryant M, Burton W, Collinson M, Hartley S, Tubeuf S, Roberts K, Sondaal AEC, Farrin AJ. Cluster randomised controlled feasibility study of HENRY: a community-based intervention aimed at reducing obesity rates in preschool children. Pilot Feasibility Stud. 2018 Jun 21;4:118. doi: 10.1186/s40814-018-0309-1. eCollection 2018. PMID 29977593
- Available data/document: Childrens Food Trust Report 2012 — http://media.childrensfoodtrust.org.uk/2015/06/CFT_Early_Years_Guide_Interactive_Sept-12.pdf — Reference 4 in citations [there-on other citations are referenced 1 citation later]